CLINICAL TRIAL: NCT05032625
Title: To Evaluate the Outcomes After Surgery for Necrotizing Soft Tissue Infections- A Prospective Longitudinal Study
Brief Title: To Evaluate the Outcomes After Surgery for Necrotizing Soft Tissue Infections
Status: Terminated | Type: Observational
Why Stopped: low accrual rate
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Rifat Latifi, The Felicien Steichen Professor and Chairman of Surgery, New York Medical College
Other Study IDs: 12943
Record Dates: First submitted 2020-08-13; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Necrotizing Soft Tissue Infection
Keywords: Necrotizing Soft Tissue Infection; Quality of life
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — Patients who undergo surgery for NSTI will be followed in hospital and for 1- year in the office. We will asses the quality of life and there functionality. This will help us in determining the predictors of poor outcome.
  Other Names: Quality of life survey

SUMMARY:
There is significant mortality associated with necrotizing soft tissue infections, it is imperative to decrease mortality and complications associated with this disease is determined. To accomplish this goal, study team will create a prospectively maintained database of all NSTI patients admitted at department of surgery. Investigators will asses the predictors of poor outcome and follow these patients for 1 year in clinic and asses the functional quality of life by incorporating 36-Item Short Form Survey (SF-36) score.

DETAILED DESCRIPTION:
RATIONALE AND BACKGROUND Necrotizing soft tissue infections (NSTIs) are severe life-threatening, rapidly-spreading, soft tissue infections of the subcutaneous tissue, fascia, or muscle caused by bacteria. Due to the rapid progression of disease, early diagnosis and treatment are crucial to a patient's survival.

Given the aggressive nature of these infections and the significant mortality associated with them, it is imperative that the optimal standard of care to decrease mortality and complications associated with this disease is determined. To accomplish this goal, study team will create a prospectively maintained database of all NSTI patients admitted at department of surgery. Investigators will follow these patients for 1 year in clinic and asses the functional quality of life by incorporating 36-Item Short Form Survey (SF-36) score. This RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It is a validated scale freely available for research to assess the quality of life after surgery.

Primary Objectives:

The short term objectives are to evaluate 30-day mortality and to establish the predictors of poor outcome. The long term objectives are to measure quality of life after NSTI.

CHARACTERISTICS OF THE STUDY POPULATION

Target Population The study population will include all patients ≥ 18 years presenting with necrotizing soft tissue infections admitted to Westchester Medical Center, who will undergo surgical management

Subject Recruitment All patients admitted with a diagnosis of NSTI who undergo or about to undergo surgery for NSTI and meet initial screening criteria will be approached by the surgeon to determine if patient will agree to participate in the research study. The PI or PI approved research personnel will explain the study to the patient or their legally authorized representative (LAR). The patient/LAR will be given adequate time to ask questions and consider participation in this study. Should the patient agree to be in the study, the PI or PI-approved research personnel will have the patient/LAR fill out the consent and HIPAA forms and they will be given a copy of both documents.

Study Design This study will be a prospective observational study. There will be no study related interventions.

Study Duration Investigators aim to enroll approximately 300 subjects between three years. Each patient will be followed for 1 year. Therefore, we expect the study will be open for at least 4 years. 3 years for enrollment and 1 year to complete the data analysis and manuscript.

DATA PROCEDURES

1. Data Collection Patients will be identified by the Department of Surgery morning report and by Emergency General Surgeons. The Emergency General Surgeons (listed at the beginning of the protocol), will notify the Department of Surgery's Clinical Research (DSCRU) unit when a patient meets study criteria. After obtaining consent, the patients will be followed up for one year. Data will be collected at the following time points: Pre-operative, Operative, Post-Operative ,2- month post-op, 4- months post-op, 8- months post-op and 1 year post-op.

Preoperative:

Demographics: age, sex, race and ethnicity Comorbidities: anemia, bleeding disorder, cancer, cardiac disease, chronic urinary tract infection, dialysis, hyperlipidemia, hypo/hyper-thyroidism, immunocompromised, prior infection, liver disease, obesity, peripheral vascular disease, renal disease, diabetes, hypertension and Transplant.

Social History: recreational drug use, tobacco and alcohol. Medications: use of anticoagulants and antiplatelets, Vitals: systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), temperature (temp), respiratory rate (resp. rate), height, weight and BMI (body mass index, Modified frailty index (Mfi) and Charleston's comorbidity index Lab reports: the lab tests that are done as standard of care during the hospital stay will be collected. The following lab values will be collected for the study only if they are available in subject's medical record: hemoglobin, hematocrit, white blood count (differential), sodium, BUN (blood urea nitrogen), lactate, pH, glucose, creatinine, platelet count, histopathology and culture for microbiology of the tissues resected during surgery, coagulation profile (PT (prothrombin time)/PTT (partial thromboplastin time) /aPTT (activated partial thromboplastin time), cultures from blood, urine, sputum, trachea, wound and peritoneal fluid will be collected as well.

Intraoperative:

Duration of surgery: start time and end time Amount and type of fluids Received: IV fluids and blood products received General: Number of drains, planned/unplanned procedures and amount of blood loss Type and number/s of surgery: Time from admission to Ist debridement (days), time from admission to 2nd debridement (days), time from admission to 3rd debridement (days, time from admission to 4th debridement (days, time from admission to 5tht debridement (days), amputation of limb (Y/N). Wound size depth (cm) (on every subsequent debridement)

Postoperative:

General: date of discharge, time of discharge, hospital length of stay, intensive care unit length of stay, (ICU LOS), ventilator days, transfer back to ICU, time of drain removal and mortality. Antibiotics (Regimen, combination, duration), hyperbaric oxygen therapy (HBOT) (Y/N), infectious disease consulted (Y/N) Complications: wound infection. Pneumonia, acute kidney injury, multi-organ dysfunction, sepsis, urinary tract infection, venous thrombosis, pulmonary embolism, adult respiratory distress syndrome Disposition: home, acute rehabilitation center, subacute rehabilitation center.

Follow up:

Investigators will follow patients for 1 year after discharge. Follow-up visits are done in the clinic after 2 weekss, 1 month, 2-months, 4-months, 8-months and 1 year of discharge. We will examine surgical site, asses pain, 36-Item Short Form Survey (SF-36) scores

The research staff will review each chart and retrieve the information included in the data collection form (please see attached). After data is collected, the research team along with the Principal Investigator along with all Co-Investigators will analyze the data.

Statistical Analysis Chi-square difference tests will be used to assess significant differences in predictors on categorical outcomes. T-tests will be used to assess mean differences in predictors on continuous outcomes. Univariable and multivariable logistic regression analyses will be conducted for outcomes such as all-cause mortality, pneumonia, sepsis, and multi-organ failure. Univariable and multivariable linear regression will be performed for hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

all patients ≥ 18 years presenting with necrotizing soft tissue infections admitted to Westchester Medical Center, who will undergo surgical management

Exclusion Criteria:

Age < 18 years.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients between 18 - 99 years of age who will undergo surgery for NSTI will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
30-day mortality. (Short term ) | 30 days
  The short term objectives are to evaluate 30-day mortality.

SECONDARY OUTCOMES:
The quality of life survey (Long Term) | 1year
  To measure quality of life survey after NSTI.

CONTACTS AND LOCATIONS:
Overall Officials: Rifat Latifi, MD, Principal Investigator — Chairman Department of Surgery
Locations (1):
- Westchester Medical center, Valhalla, New York, United States